CLINICAL TRIAL: NCT02878759
Title: Wristbot: A Novel Device for the Assessment of Proprioceptive Deficits After Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/00502
Record Dates: First submitted 2016-08-17; First posted 2016-08-25 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Prospective single arm intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wristbot (Experimental): WristBot will be used as diagnostic tool to evaluate the novel technology and the associated protocol for proprioception quantification during rehabilitation. The main objective is to provide clinicians with a reliable instrument able to overcome the limitations in proprioceptive measurement by current clinical methodologies.
  Interventions: Device: Wristbot

INTERVENTIONS:
Device: Wristbot — The proposed technology comprises a hardware device with four motors that can apply torques to the human wrist about its three degrees of freedom (i.e. axes of rotation: wrist flexion/extension,abduction/adduction and forearm pronation/supination). This allows for guided and controlled movements of the wrist by delivering assistive, resistive, perturbation or no forces (patient actively moves the wrist). It contains a set of specialized software modules that a) allow for the objective, psychophysical assessment of sensory dysfunction in patients, and b) provide specialized training modules designed to improve sensory and motor functions of the wrist.

SUMMARY:
The WristBot constitutes a comprehensive, integrated robotic system for the early diagnosis and rehabilitation of sensory and fine motor dysfunction to neurological or orthopedic disease.

DETAILED DESCRIPTION:
The WristBot constitutes a comprehensive, integrated robotic system for the early diagnosis and rehabilitation of sensory and fine motor dysfunction to neurological or orthopedic disease. It has been validated in three clinical trials, including orthopaedic patients, Parkinsons disease and 9 chronic stroke patients. Its unique feature uses adaptive, progressive robot-aided therapy to achieve intensive, task specific wrist movements.

In the context of the proposed project we will target the stroke population. Integration refers here to the system's ability to perform the assessment of proprioceptive status and proprioceptive training in a single device. The scope of the current project is investigating the efficacy of the proprioceptive assessment of the WristBot and correlating the result throughout the rehabilitation protocol. The proposed technology comprises a hardware device with four motors that can apply torques to the human wrist about its three degrees of freedom (i.e. axes of rotation: wrist flexion/extension,abduction/adduction and forearm pronation/supination). This allows for guided and controlled movements of the wrist by delivering assistive, resistive, perturbation or no forces (patient actively moves the wrist). It contains a set of specialized software modules that a) allow for the objective, psychophysical assessment of sensory dysfunction in patients, and b) provide specialized training modules designed to improve sensory and motor functions of the wrist.

ELIGIBILITY:
Inclusion Criteria:

* First clinical stroke (ischaemic or haemorrhagic) diagnosed by brain imaging CT or MRI
* Age 21 years to 85 years, both males and females.
* < 90 days of stroke on admission to rehabilitation
* Presence of either motor and /or sensory deficit detected by clinical examination.
* Ability to understand simple instructions.
* Ability to give own consent.
* Ability to sit supported in a chair for 60 minutes with appropriate rest breaks.

Exclusion Criteria:

* Non stroke -related causes of motor/sensory deficits
* Tetraplegia or tetraparesis
* Known diagnosis of cervical myelopathy, lower motor neuron weakness (Post polio, brachial plexopathy, peripheral neuropathy (Diabetic, carpel tunnel syndrome, B12 deficiency)
* Concomitant orthopaedic condition limiting wrist range of motion: active arm/wrist fractures, fixed contractures of the wrist joint, wrist joint arthritis, wrist fusion.
* Arm or wrist joint pain (Visual Analogue scale VAS >5/10) or instability
* Severe hemispatial neglect.
* Significant wrist spasticity with modified Ashworth Scale score 2 and above.
* Life expectancy <6 months, end stage renal or liver disease, terminal cancer.
* Pregnancy and lactation in female patients.
* Postural hypotension on sitting up
* Active skin conditions over wrist joint area which could be worsened by robotic fit (e.g. severe eczema, burns)

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Fugyl Meyer assessment motor assessment score (FMA 0-66) | 2 years
  To assess motor impairment of affected upper limb
Wolf Motor Function Test for affected limb (WMFT), | 2 years
  To assess motor impairment of affected upper limb
Nine hole peg test (in seconds) | 2 years
  brief, standardized, quantitative test of upper extremity function
Functional Independence Measure | 2 years
  Test of upper limb function
Modified Ashworth Scale | 2 years
  Test of muscle spasticity for upper limb
standardised somatosensory deficit index | 2 years
  Sensory assessment of upper limb
Visual Analogue scale | 2 years
  Scale to assess pain

CONTACTS AND LOCATIONS:
Overall Officials: Karen SG Chua, MBBS/MRCP, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital CART 5B, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No